CLINICAL TRIAL: NCT00164957
Title: The Effect of Continuous vs Enteral Pump Feeding in Aspiration in Tube Fed Patients
Brief Title: The Effect of Continuous Versus Enteral Pump Feeding in Aspiration in Tube Fed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RCT-pumpfeeding
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration

INTERVENTIONS:
Device: continuous pump feeding
Other: intermittent bolus feeding

SUMMARY:
Background:

Tube feeding had been found to be a cause of aspiration pneumonia. Continuous pump feeding at slower rates as compared to bolus feeding may be less associated with aspiration pneumonia.

Methods:

Randomized controlled trial

Subjects:

Patients expected to remain on tube feeding for 4 or more weeks

Outcomes:

1) pneumonia, 2) mortality

DETAILED DESCRIPTION:
Eligible subjects are randomized into 2 groups by random numbers generated by a computer programme: intermittent bolus feeding versus continuous feeding via a delivery pump.

Baseline Assessment:

Clinical details including background medical diagnoses, indications for enteral feeding, functional status and baseline CXR findings are recorded.

Tube Feeding Regime:

The choice of feeding formula and feeding volume will be guided by 2 dietitians collaborating in this study. Giving sets for continuous pump feeding are changed everyday.

Pump feeding is defined at delivery rate <60ml/hr. In order to avoid interfering with rehabilitative activities, pump feeding can be discontinued for no more than eight hours during the day. Bolus feeding is defined as no more than 400ml/hr, 4 to 5 times per day.

All subjects are reviewed to monitor complications arising from enteral feeding. Free pump feeding sets will be provided for an extra 2 weeks for pump feeding group subjects discharged before the end of the trial. All subjects discharged prior to the end of trial will be contacted regularly by a research assistant until completion or outcome is reached.

Outcome Pneumonia is diagnosed in the presence of 2 major clinical signs: increased sputum production and pneumonic changes in the CXR (according to radiologist report), or in the presence of one major sign and 2 of the following minor clinical signs: raised or depressed white cell count, hypoxia at room air (PaO2 <92%) and body temperature greater than 38%. When the criteria for pneumonia are fulfilled, the trial will be terminated.

All the subjects are followed up for four weeks or until outcome is reached (i.e. pneumonia). Mode of tube feeding on discharge will be decided by the attending physicians, patients and family members.

ELIGIBILITY:
Inclusion Criteria:

* patients likely to need tube feeding for another 4 weeks

Exclusion Criteria:

* Patients already on pump feeding.
* Active sepsis: fever, abnormal white cell count
* CXR shadowing
* Chronic hypoxia (O2 saturation <92% on room air)
* Patients who have a history of recurrent self-extubation.
* Short life expectancy (within weeks)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2002-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
pneumonia | within 4 weeks

SECONDARY OUTCOMES:
mortality | within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy CY Kwok, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, China